CLINICAL TRIAL: NCT03031184
Title: A Pragmatic, Multi Centre, Double-blind, Placebo Controlled Randomised Trial to Assess the Safety, Clinical and Cost Effectiveness of Mirtazapine in Patients With Alzheimer's Disease (AD) and Agitated Behaviours
Brief Title: Study of Mirtazapine for Agitation in Dementia
Acronym: SYMBAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sussex (Other)
Collaborators: Norwich Clinical Trials Unit (Unknown); University of East Anglia (Other); University of Cambridge (Other); University College, London (Other); London School of Economics and Political Science (Other); University of Manchester (Other); University of Newcastle Upon-Tyne (Other); Birmingham and Solihull Mental Health NHS Foundation Trust (Other); Alzheimer's Society (Other); The Centre for Dementia Studies, Brighton and Sussex Medical School and SPFT (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15/SC/0606
Record Dates: First submitted 2017-01-03; First posted 2017-01-25 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Dementia
Keywords: Agitation; Agitated behaviours; Alzheimer's Disease
MeSH Terms: conditions — Dementia; Psychomotor Agitation; Alzheimer Disease | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirtazapine (Experimental): 15mg of Mirtazapine over encapsulated to produce a blinded product that looks identical to the other arms. Starting dose is one capsule per day, escalating to 2 capsules per day after 2 weeks if no side effects and up to 3 capsules per day after 4 weeks.
  Interventions: Drug: Mirtazapine
- Placebo (Placebo Comparator): Lactose powder encapsulated to produce a blinded product that looks identical to the other arms. Starting dose is one capsule per day, escalating to 2 capsules per day after 2 weeks if no side effects and up to 3 capsules per day after 4 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mirtazapine
  Arms: Mirtazapine
Other: Placebo
  Other Names: Dummy pill
  Arms: Placebo

SUMMARY:
This clinical trial evaluates whether Mirtazapine is more effective than placebo in treating agitation in people with dementia. The trial will assess the safety, clinical and cost effectiveness of the treatment. Participants will be randomised to receive either Mirtazapine or placebo for 12 weeks and will be followed up for up to one year, in this blinded trial.

DETAILED DESCRIPTION:
Patient-centred care, without the use of medicines is offered as a first course of treatment for agitation in dementia. However, there is a need for second line treatments when these fail, at the moment antipsychotics are commonly prescribed, as very little research has been done in to safer alternative treatments.

There are medicines available to treat agitation and/or aggression in dementia, but it is not clear which treatments work best.

This research study has been designed to help answer this, by comparing a which is currently prescribed for depression, Mirtazapine, with placebo (a tablet designed to look like a medicine but that has no active medicine in it) to see if Mirtazapine is suitable for treating agitation in dementia.

If participants and their family/carers agree to take part in this study, participants will be prescribed treatment for 12 weeks. Participants will then be followed up for 1 year after, with assessment sessions at 26 and 52 weeks.

Participants taking part in this study will be randomly allocated to a treatment group (selected to their treatment group by chance). The study is blinded, so this means the participant's doctor and the research team will not know which treatment the participant has been taking until after the study has ended. This is necessary so that the trial is a fair test of which treatment works best, however it is possible to find out which medicine they are taking in the event of a medical emergency.

The study is entirely voluntary and all participants wishing to join the study must complete an informed consent form (or if they lack capacity the participant's representative may do so on their behalf). Each participant must also have a nominated carer who consents to being questioned on aspects of the participant's dementia/care and their own experiences in caring for the participant.

The investigators are aiming to recruit 222 patients to the study in total from around 20 different regions across the UK.

The study was originally designed to included a second medication, called Carbamazepine, to also look at whether it would work and be safe and cost effective in agitation in dementia. Challenges in recruitment in this population resulted in the funder requesting that the available data was reviewed to July 2018, to see whether one of the arms (Mirtazapine or Carbamazepine) should be discontinued in terms of future recruitment. The independent data monitoring committee compared blinded data from both groups against placebo data and concluded that on the basis of efficacy and safety, the group, which when unblinded was found to be Carbamazepine, should be dropped. Some limited analysis will still be completed for all data collected in the Carbamazepine group, but the trial will continue now only randomising participants to Mirtazapine or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of probable or possible Alzheimer's Disease using National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria (McKhann et Al, 1984)
* a diagnosis of co-existing agitated behaviours
* evidence that the agitated behaviours have not responded to management according to the AS/DH algorithm (AS/DH, 2011)
* An assessment of Cohen Mansfield Agitation Inventory (CMAI; Cohen-Mansfield et al, 1989, Long form) score of 45 or greater
* Written informed consent to enter and be randomised into the trial
* Availability of a suitable informant (consenting identifiable family carer or paid carer) to provide information on carer-completed outcome measures and who consents to take part in the trial.

Exclusion Criteria:

* Current treatment with antidepressants (including MAOIs) or antipsychotics. Normal clinical practice should be followed, with an appropriate washout period before trial drug administration. For MAOIs this should be least two weeks.
* Contraindications to the administration of mirtazapine as per the current SmPC
* Patients with second degree atrioventricular block (patients with third degree heart block, with a pace maker fitted, may be included at PI discretion)
* Cases too critical for randomisation (ie where there is a suicide risk or where the patient presents a risk of harm to others)
* Female subjects under the age of 55 of childbearing potential, defined as follows: postmenopausal females who have not had at least 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhoea with serum FSH>40mIU/ml or females who have not had a hysterectomy or bilateral oophorectomy at least 6 weeks prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Cohen Mansfield Agitation Inventory (CMAI) score (Long Form, 29 questions) | Baseline, 6 weeks, 12 weeks
  Measured at baseline, 6 and 12 weeks, it is the difference in the score at 12 weeks that is the primary outcome. The questions are asked of the person with dementia's carer

CONTACTS AND LOCATIONS:
Overall Officials: Sube Banerjee, Professor, Principal Investigator — Brighton and Sussex Medical School
Locations (1):
- Sube Banerjee, Brighton, Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during the current study will be available upon request from Prof Sube Banerjee sube.banerjee@plymouth.ac.uk once the trial follow-up and analyses are completed, the likely date for this is October 2022.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After analysis by the study team is complete, likely from October 2022. The above documents are already available
Access Criteria: By email request to Prof Sube Banerjee sube.banerjee@plymouth.ac.uk

REFERENCES:
- [Derived] Banerjee S, Farina N, Henderson C, High J, Stirling S, Shepstone L, Fountain J, Ballard C, Bentham P, Burns A, Fox C, Francis P, Howard R, Knapp M, Leroi I, Livingston G, Nilforooshan R, Nurock S, O'Brien J, Price A, Thomas AJ, Swart AM, Telling T, Tabet N. A pragmatic, multicentre, double-blind, placebo-controlled randomised trial to assess the safety, clinical and cost-effectiveness of mirtazapine and carbamazepine in people with Alzheimer's disease and agitated behaviours: the HTA-SYMBAD trial. Health Technol Assess. 2023 Oct;27(23):1-108. doi: 10.3310/VPDT7105. PMID 37929672
- [Derived] Banerjee S, High J, Stirling S, Shepstone L, Swart AM, Telling T, Henderson C, Ballard C, Bentham P, Burns A, Farina N, Fox C, Francis P, Howard R, Knapp M, Leroi I, Livingston G, Nilforooshan R, Nurock S, O'Brien J, Price A, Thomas AJ, Tabet N. Study of mirtazapine for agitated behaviours in dementia (SYMBAD): a randomised, double-blind, placebo-controlled trial. Lancet. 2021 Oct 23;398(10310):1487-1497. doi: 10.1016/S0140-6736(21)01210-1. PMID 34688369